CLINICAL TRIAL: NCT06137157
Title: A Randomized, Double-Blind, Vehicle-Controlled, First-in-Human Safety, Tolerability and Proof-of-Concept Study of Topical ATR12-351 in Adults With Netherton Syndrome
Brief Title: Evaluation of Topical ATR12-351 in Adults With Netherton Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Azitra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTH201
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Netherton Syndrome
Keywords: Ichthyosis; Netherton syndrome; Skin disease; ichthyosis linearis circumflexa
MeSH Terms: conditions — Netherton Syndrome; Ichthyosis; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Intrapatient, randomized controlled study: ATR12-351 will be applied to skin lesions on one side of the body, while the vehicle control will be applied to similar lesion on the other side of the body twice daily for 2 weeks. Each patient is randomized to receive ATR12-351 on either the left or right side.
Masking Description: Patients, investigators, and assessors will be masked as to whether patients received ATR12-351 on the right or left side of the body.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Internal controlled arm (Experimental): ATR12-351 on left side of body, vehicle on right side of body in one group; vehicle on left side of body, ATR12-351 on right side of body.
  Interventions: Drug: ATR12-351

INTERVENTIONS:
Drug: ATR12-351 — Topical ointment containing ATR12-351, a LEKTI-secreting strain of S. epidermidis
  Other Names: ATR-12

SUMMARY:
The objectives of this clinical trial are to evaluate the safety and tolerability of topically applied ATR12-351, to understand what the body does to ATR12-351, and to observe treatment benefits of the drug in approximately 12 adult patients with Netherton Syndrome (NS). ATR12-351 will be applied to skin lesions on one side of the body, while the vehicle control will be applied to similar lesion on the other side of the body twice daily for 2 weeks.

DETAILED DESCRIPTION:
Netherton syndrome (NS) is a rare but severe autosomal recessive disease that affects the skin, hair, and immune system. NS presents at birth with red skin covered by fine scales, a specific hair shaft abnormality ("bamboo hair"), atopic lesions, and elevated systemic immunoglobulin E (IgE) levels. Patients often develop allergies and asthma, and the unfortunate prognosis for infants with NS is poor, with 10% mortality in the first 6 months of life and recurrent infections. There are no FDA-approved treatment options for NS. NS is caused by mutations in in the SPINK5 gene encoding the serine protease inhibitor lymphoepithelial Kazal-type related inhibitor (LEKTI). Absence of LEKTI causes unregulated activity of proteases in the kallikrein subfamily, causing excessive desquamation of skin.

ATR12-351 is a topical ointment containing a lyophilized version of a live biotherapeutic product (LBP), Staphylococcus epidermidis (SE) strain designated SE351. This strain has been modified to be auxotrophic and to express recombinant human LEKTI protein (rhLEKTI). ATR12-351 is intended to address the underlying cause of NS by replacing deficient/dysfunctional LEKTI. The treatment consists of applying ATR12-351 to affected areas, where rhLEKTI produced by ATR12-351 will counter the dysregulated skin serine protease activity observed in NS patients.

This first-in-human study is a randomized, double-blind, vehicle-controlled clinical study to assess the safety, tolerability, and pharmacokinetics (PK) of topical ATR12-351 in approximately 12 adult Netherton syndrome patients who will serve as their own control. This study will include a 14-day treatment period to investigate the safety and tolerability of ATR12-351 applied to the skin and will be followed a total of 84 days for safety. The results of this first-in-human clinical study will establish safety and tolerability as well as initial efficacy of ATR12-351 application in Netherton syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Confirmed mutation of the serine protease inhibitor of Kazal type 5 (SPINK5) gene
* Involvement of ≥20% of body surface area with skin changes consistent with Netherton syndrome

Exclusion Criteria:

* Use of biologic therapies, antibiotics, antihistamines, corticosteroids, retinoids, disease-modifying antirheumatic drugs (DMARDs), immunosuppressive agents, phosphodiesterase-4 (PDE4) inhibitors, topical calcineurin inhibitors, or topical Janus kinase (JAK) inhibitors
* Open wounds or extensive areas of excoriation precluding identification of appropriate application sites in the Investigator's judgment
* Concurrent involvement in any other clinical study/expanded access program with an investigational drug or device or has participated in a clinical study within 30 days prior to the screening visit
* Residing with an immunocompromised person in the same dwelling from the baseline visit through 2 weeks after the treatment period
* History of ultraviolet phototherapy within the planned treatment area 4 weeks prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 84 days
  Incidence, severity, seriousness and relatedness of all treatment-emergent adverse events

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) | 42 days
  Visual assessment of the overall severity of skin disease severity at each application site, using a 5-point scale (0, clear; 1, almost clear/minimal; 2, mild; 3, moderate; 4, severe). Higher scores indicate greater severity.
Patient's Global Assessment (PGA) | 42 days
  Visual assessment of the overall severity of skin disease severity at each application site, using a 5-point scale (0, clear; 1, almost clear/minimal; 2, mild; 3, moderate; 4, severe). Higher scores indicate greater severity.
NS-modified SCORAD | 42 days
  The investigator's objective assessment of the severity (peeling, scaling, lichenification, erythema, papules) and extent (surface of affected skin areas) of skin disease at each application site is combined with patient's subjective scores (pain and pruritus). Higher scores indicate greater severity with a maximum of 100 points possible.
Pharmacokinetics: plasma concentration | 42 days
  Concentration (ng/mL) of rhLEKTI in the plasma following topical application.
Pharmacokinetics: skin concentration (Cmax skin) | 42 days
  Concentration of rhLEKTI in the skin (pmol/cm2), measured by tape stripping, following topical application.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, MD, Study Director — Azitra Inc.
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No